CLINICAL TRIAL: NCT04981691
Title: An Open, Single-center, Exploratory Clinical Trial to Evaluate the Safety and Efficacy of mRNA CAR-mesothelin T Cells in Patients With Advanced Refractory Solid Tumors
Brief Title: Anti-mesothelin CAR-T Cells With Advanced Refractory Solid Tumors
Acronym: Amaretto
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Ruijin Hospital (Other)
Collaborators: UTC Therapeutics Inc. (Industry)
Responsible Party: Principal Investigator, Jun Zhang, Chief of Department of Oncology, Ruijin Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Amaretto
Record Dates: First submitted 2021-07-07; First posted 2021-07-29 (Actual); Last update posted 2021-09-17 (Actual); Status verified 2021-09

CONDITIONS: Refractory Malignant Solid Neoplasm
Keywords: Mesothelin; Refractory Solid Tumors; Chimeric Antigen Receptor T-Cell; Phase I clinical trial

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- anti-MESO CAR-T cells (Experimental): The subjects in this arm will receive Cyclophosphamide 300mg/m2/d and Fludarabine 30mg/m2/d from day-4 to day-2. Subjects will be treated with six administrations of anti-MESO CAR-T cells three times weekly (Monday-Wednesday-Friday) for two weeks. In the first week, total 1×109 or 3×109 will be infused, the second week is to plan three times consecutive infusions of 1x109 or 3×109 anti-MESO CAR-T cells each time.
  Subjects will be enrolled serially. For subject safety, the preceding subject must have completed therapy and be 28 days from their last infusion before the next subject can be treated.
  Interventions:
  * Drug: anti-MESO CAR-T cells
  * Drug: Fludarabine
  * Drug: Cyclophosphamide
  Interventions: Biological: anti-MESO CAR T cells

INTERVENTIONS:
Biological: anti-MESO CAR T cells — Autologous genetically modified anti-MESO CAR T cells

SUMMARY:
The goal of this clinical trial is to study the safety, efficacy, and pharmacokinetics of mRNA-engineered anti-Mesothelin (MESO) Chimeric Antigen Receptor T-Cell (CAR-T cells) therapy in patients with mesothelin expression-positive, advanced solid tumors that have failed at least first-line or second-line therapy.

DETAILED DESCRIPTION:
This phase I study is being conducted to establish safety, pharmacokinetics, and preliminary efficacy of intravenous (IV) mRNA electroporated fully-humanized anti-MESO re-directed autologous T cell administration in patients with chemotherapy-refractory metastatic solid tumors.

The study will adopt the "3+3" dose escalation design exploring two doses of 1×109 and 3×109. The administration is planned to infuse 3 times a week for 2 consecutive weeks.

• The subjects will receive a total dose of 1x109 RNA transduced anti-MESO CAR-T cells in the first week, following lymphodepleting chemotherapy with cyclophosphamide 300 mg/m2/day and fludarabine 30 mg/m2/day given over 3 days by intravenous infusion. If there is no obvious dose-limiting toxicity (DLT) after the first week of infusion, three times consecutive infusions of 1x109 anti-MESO CAR-T cells each time is planned in the second week. Each subject needs to be observed for at least 2 weeks (14 days) after completing the last infusion. Lymphodepleting chemotherapy will not be repeated prior to additional infusions of anti-MESO CAR-T cells.

ELIGIBILITY:
Inclusion Criteria:

1. Ability to understand and the willingness to provide written informed consent.
2. Advanced pancreatic cancer, ovarian cancer, malignant mesothelioma, gastric cancer, bowel cancer, etc., diagnosed by histopathological or cytological examination, but not limited to subjects with various advanced solid tumors.
3. IHC test showed Mesothelin positive expression at least 1+ in tumor tissue
4. Age no less than 18 years.
5. Life expectancy greater than 3 months.
6. According to the RECIST (Response Evaluation Criteria in Solid Tumors) standard, there must be measurable lesions.
7. Evidence of metastatic disease and failure of at least 1 prior chemotherapy for metastatic disease. During the last treatment or after the treatment, the disease progressed and was confirmed (the investigator judged according to the RECIST 1.1 standard).
8. Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1 during the screening period and before apheresis.
9. Adequate liver/bone marrow function.
10. Female subjects must meet the following conditions: infertility or fertility and use high-efficiency contraceptive measures.
11. Male subjects agree to use approved contraceptive methods (e.g. birth control pills, barrier device, intrauterine device, abstinence) during the study and for 3 months following the last dose of the study cell infusion. Moreover, all men are absolutely prohibited from donating sperm within 1 year after receiving the last study treatment infusion.

Exclusion Criteria:

1. Participated in any other trial in which receipt of an investigational study drug occurred within 28 days prior to entry into the study.
2. Received any anticancer medication in the 2 weeks prior to receiving their first dose of study treatment, including but not limited to surgery, systemic chemotherapy, radiotherapy, intervention, etc.
3. Uncontrolled thyroid dysfunction (serum thyroid hormone determination TT4, TT3, FT3, FT4, and serum thyroid-stimulating hormone TSH) are not suitable for enrolling in the study;
4. Pregnant or breastfeeding female, or not willing to take contraception measures during the study.
5. Any uncontrollable active infection, including but not limited to active tuberculosis; HBV infection (including HBsAg positive, or HBcAb positive and HBV DNA positive); HIV, syphilis, hepatitis C positive or suffering from other fatal viruses, Bacterial disease
6. Administrated with steroids (5 mg/day or more dexamethasone, or equivalent hormone drugs) within the past two weeks;
7. Other uncontrolled diseases may cause abnormal death of the patient;
8. Active autoimmune disease (including but not limited to: systemic lupus erythematosus, Sjogren's syndrome, rheumatoid arthritis, psoriasis, multiple sclerosis, inflammatory bowel disease, etc.) requiring immunosuppressive therapy within the past 4 weeks.
9. Previously allergic to immunotherapy, tocilizumab, cyclophosphamide, fludarabine, and other related drugs, previous history of severe allergies, to research product excipients (such as human serum albumin, DMSO, and dextran 40 ); people who have a history of penicillin allergy and have a positive skin test at the time of screening.
10. Congestive heart failure, uncontrolled cardiac arrhythmia, etc.
11. Uncontrollable massive ascites, that cannot be drained by standard methods;
12. Intestinal obstruction or CT suggesting omental cake-like peritoneal metastasis, or repeated uncontrollable incomplete intestinal obstruction.
13. Have received any genetic engineering modified T cell therapy (including CAR T, TCR T cell).
14. Uncontrolled brain metastasis or mental illness.
15. Suffered from other uncured malignant tumors within the past 3 years or at the same time.
16. The blood oxygen saturation ≤95% at the time of screening and before apheresis.
17. Can't be followed up or obey protocol.
18. The investigator believes that it is not appropriate to participate in the trial.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2021-10-01 (Estimated); Primary Completion 2022-01-09 (Estimated); Study Completion 2022-07-09 (Estimated)

PRIMARY OUTCOMES:
TEAEs | 4 weeks after the last infusion
  Incidence of Treatment Emergent Adverse Event
TRAEs | 4 weeks after the last infusion
  Incidence of Treatment Related Adverse Events
SIAEs and SAEs | 4 weeks after the last infusion
  Incidence of AEs of Special Interest and Serious Adverse Events
DLTs | 4 weeks after the last infusion
  Incidence of dose-limiting toxicities

SECONDARY OUTCOMES:
TEAEs,TRAEs, SIAEs and SAEs | 12 weeks after the last infusion
  Incidence of Treatment Emergent Adverse Event, Treatment Related adverse events, AEs of special interest and serious adverse events
ORR by IR | 12 weeks after the last infusion
  Objective response rate based on investigator's evaluation
ORR by IRC | 12 weeks after the last infusion
  ORR based on independent review committee evaluation
DCR by IR | 12 weeks after the last infusion
  Disease control rate based on the investigator's evaluation
DCR by IRC | 12 weeks after the last infusion
  DCR based on IRC evaluation
DOR by IR | 12 weeks after the last infusion
  Duration of Remission based on the investigator's evaluation
TTR by IR | 12 weeks after the last infusion
  Time to remission based on the investigator's evaluation
PFS by IR | 24 weeks after the last infusion
  Progression-free survival (PFS) based on the investigator's evaluation
PFS by IRC | 24 weeks after the last infusion
  PFS based on IRC evaluation
OS | 52 weeks after the last infusion
  Overall survival
QOL | 12 weeks after the last infusion
  According to the EUROPEAN Organization for Research and Treatment of Cancer, Eortc, Quality of Life QuestionNare-Core 3, QOQ-C30), ERTC QLQ-C30, evaluated subject's quality of life.
Cmax | 4 weeks after the last infusion
  the highest concentration (Cmax) of anti-human MESO T cells in the peripheral blood after CAR T cell infusion
AUC | 4 weeks after the last infusion
  the area under the curve of 28 days of anti-human MESO T cells in the peripheral blood after CAR T cell infusion
HACA | 4 weeks after the last infusion
  Positive rate of Human Anti-CAR Antibodies after CAR T cell infusion

OTHER OUTCOMES:
mesothelin expression and efficacy | 12 weeks after the last infusion
  Immunohistochemical method to detect the expression of mesothelin, CT or magnetic resonance image（MRI） evaluation efficacy, statistical method (SPSS 24.0) to assess the correlation between mesothelin expression level and efficacy

CONTACTS AND LOCATIONS:
Overall Officials: Jun Zhang, MD, PhD, Principal Investigator — Ruijin Hospital
Locations (1):
- Department of Oncology, Ruijin Hospital, Shanghai, China

IPD SHARING:
Plan to Share IPD: No